CLINICAL TRIAL: NCT04727164
Title: An Open Phase I Study to Evaluate the Safety, Tolerability, PK / PD, and Initial Efficacy of HBM4003 in Combination With Toripalimab in Patients With Advanced Melanoma and Other Solid Tumors
Brief Title: Study Investigating Safety,Tolerability,Pharmacokinetics and Antitumor Activities of HBM4003 Combine With Toripalimab
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Harbour BioMed (Guangzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4003.2
Record Dates: First submitted 2020-12-08; First posted 2021-01-27 (Actual); Last update posted 2021-01-29 (Actual); Status verified 2021-01

CONDITIONS: Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HBM4003+Toripalimap (Experimental): HBM4003 combined with toripalimab in patients with advanced melanoma and other solid tumors
  Interventions: Drug: HBM4003 and Triprilimab

INTERVENTIONS:
Drug: HBM4003 and Triprilimab — Subjects will be treated with HBM4003 on Day 1 Cycle 1 and be treated with HBM4003 and Triprilimab during each 21-day cycles from Cycle 2 in part 1.Subjects will be treated with HBM4003 and Triprilimab on Day 1 during each 21-day cycle in part 2.
  Other Names: HBM4003

SUMMARY:
HBM4003 in combination with Toripalimab. The expected duration of treatment for each subject will vary according to the number of cycles completed; the number of cycles will depend on whether the subject benefits from the treatment. The study consists of a 4-week screening period, a 21-day treatment cycle (repeatable, depending on the presence/absence of clinical benefit), EOT visit after discontinuation of treatment, and 2 follow-up visits 28 days (± 2 days) and 84 days (± 5 days) after the last study medication.

DETAILED DESCRIPTION:
An open-label Phase 1 study to evaluate the safety, tolerability, PK/PD and preliminary efficacy of HBM4003 combined with toripalimab in patients with advanced melanoma and other solid tumors.

The study is composed of two part, part 1 will be approximately 31subjects and Part 2 will be approximately 30 subjects.

ELIGIBILITY:
Main inclusion/exclusion criteria:

Main inclusion criteria

1. Males or females aged ≥ 18 years at the time of signing the informed consent form. For Part 1 of this study, the subjects should be ≤ 75 years of age.
2. For Part 1 of the study, patients histopathologically diagnosed with advanced or recurrent solid tumors
3. For Part 2 of the study, patients with locally advanced or metastatic melanoma who had been pathologically confirmed and could not be surgically removed were enrolled.
4. Subjects must be able to provide fresh or archived tumor tissues .
5. Patients whose estimated survival time is more than 3 months.
6. Patients with at least one measurable lesion at baseline according to RECIST (Version 1.1).
7. Patients with Eastern Cooperative Oncology Group (ECOG) performance status score ≤ 1.
8. Patients whose organ function must meet the study requirements:
9. Every woman or man with potential fertility needs to use an effective contraceptive method.

Main exclusion criteria

1. Patients who are simultaneously participating in another clinical study, unless the study is an observational (non-interventional) clinical study or the patient is already in the survival follow-up period of the interventional study.
2. Patients with a history of severe allergic diseases, a history of severe drug allergies, and known or suspected allergy to macromolecular protein preparations or HBM4003 excipients or toripalimab excipients.
3. Previous and concomitant drugs or treatments to be excluded like CTLA4, PD-1,PD-L1.
4. Insufficient recovery from previous treatments:
5. Diseases that may affect the efficacy and safety of the investigational product.
6. A history of other malignant diseases within 5 years before the first dose.
7. Symptomatic, active, or urgent treatment-requiring central nervous system (CNS) metastasis with imaging evidence (based on CT or MRI assessment).
8. Subjects with pleural effusion, pericardial effusion, or ascites
9. Subjects who the investigator believes may have other factors that will affect the efficacy or safety evaluation of this study (e.g., mental disorders, alcoholism, drug use, etc.).
10. Women who are pregnant or breastfeeding, or who plan to become pregnant during the study period and within 3 months after the last administration of the investigational product.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Estimated)
Dates: Start 2021-02-28 (Estimated); Primary Completion 2023-11 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Prat 1 :MTD | approximate 42 days
  The maximum tolerated dose (MTD) of HBM4003 combined with toripalimab
Prat 1 :RP2D | approximate 42 days
  Recommended Phase 2 dose (RP2D) of HBM4003 combined with toripalimab
Part 1:Number of subjects with DLT in each dose group within 2 cycles (42 days) after the first trial administration | approximate 42 days
  DLT observation period was defined as two treatment cycles with a total of 42 days,including 21 days in the first cycle (HBM4003 single drug treatment cycle) and 21 days in the second cycle (HBM4003 combined with triprilimab treatment cycle).
Part 2:ORR | maximum 3 years
  Proportion of patients with complete response (CR) and partial response (PR)

SECONDARY OUTCOMES:
Part 1:ORR | maximum 3 years
  Proportion of patients with complete response (CR) and partial response (PR)
Part 1:Disease Control Rate，DCR | maximum 3 years
  Including complete response (CR),partial response (PR) and disease stability (SD)
Part 1:Duration of Response, DOR | maximum 3 years
  Calculate the duration from the first confirmed CR or PR to the date of disease progression or death (for any reason)
Part 1:Duration of Disease Control, DDC | maximum 3 years
  For subjects with Cr, PR or SD, the duration from the time of initial administration to the date of disease progression or death (for any reason) was calculated
Cmax (Maximum serum concentration) | maximum 3 years
  Cmax
Tmax (Time to reach maximum serum concentration) | maximum 3 years
  Tmax
AUC0-last | maximum 3 years
  AUC0-last
AUC0-tau (Area under the serum concentration versus time curve from time zero to the dosing interval tau | maximum 3 years
  AUC0-tau
The immunogenicity of HBM4003 and Triprilimab | maximum 3 years
  Including the incidence of ADA positive. For ADA positive patients, the incidence of neutralizing antibody (NAB) was analyzed.
Part 2:DCR | maximum 3 years
  Proportion of patients with CR, PR and SD
Part 2:DOR | maximum 3 years
  Calculate the duration from the first confirmed CR or PR to the date of disease progression or death (for any reason)
Part 2:DDC | maximum 3 years
  For subjects with Cr, PR or SD, the duration from the time of initial administration to the date of disease progression or death (for any reason) was calculated
Prat 2:OS | maximum 3 years
  The length of time from the beginning of treatment to the death of the subject (for any reason)
Part 2:PFS | maximum 3 years
  The length of time from the beginning of treatment to the onset of disease progression or (for any reason) death;
Prat 2:The immunogenicity of HBM4003 and Triprilimab | maximum 3 years
  Including the incidence of ADA positive. For ADA positive patients, the incidence of neutralizing antibody (NAB) was analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: JUN GUO, DOCTOR, Principal Investigator — Peking University Cancer Hospital & Institute

REFERENCES:
- [Derived] Tang B, Chen Y, Jiang Y, Fang M, Gao Q, Ren X, Yao L, Huang G, Chen J, Zhang X, Li R, Zhao S, Gao M, Luo R, Qi M, Li F, Zheng F, Lee M, Tao X, Duan R, Guo J, Chi Z, Cui C. Toripalimab in combination with HBM4003, an anti-CTLA-4 heavy chain-only antibody, in advanced melanoma and other solid tumors: an open-label phase I trial. J Immunother Cancer. 2024 Oct 4;12(10):e009662. doi: 10.1136/jitc-2024-009662. PMID 39366752